CLINICAL TRIAL: NCT05760287
Title: Echocardiographic Characterization of Cardiac Amyloidosis: an Observational Study
Brief Title: Echocardiographic Characterization of Cardiac Amyloidosis
Acronym: Echo-AMY
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5308
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Amyloidosis
Keywords: echocardiography; left ventricle
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a mono-center observational ambispective study in which patients with cardiac amyloidosis evaluated at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Rome, Italy) will be enrolled.

The primary aim is to investigate echocardiographic findings, particularly using advanced echocardiographic techniques, such as two- and three-dimensional speckle-tracking analysis, that may be helpful in the differential diagnosis between cardiac amyloidosis and other cardiomyopathies with hypertrophic phenotype.

Secondary aims are: 1) to evaluate the reversibility of myocardial damage, assessed by echocardiography, in response to a newly available specific treatment for patients with transthyretin-related cardiac amyloidosis (tafamidis) and its correlation with the clinical response 2) to investigate potential novel echocardiographic predictors of adverse cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients with cardiac amyloidosis, defined according to the recommendations provided by the working group of the european society of cardiology, with clinical, electrocardiographic ed echocardiographic data and with at least one follow-up visit.

Exclusion Criteria:

* missing data
* decline to the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the retrospective phase, patients with cardiac amyloidosis evaluated at the Fondazione Policlinico Agostino Gemelli between January 2020 and November 2022 will be enrolled.
  In the prospective phase, patients with the same features evaluated between December 2022 and December 2028.
Sampling Method: Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2030-12-02 (Estimated); Study Completion 2031-02-02 (Estimated)

PRIMARY OUTCOMES:
changes in echocardiographic parameters (in patients receiving or not specific treatment) | 6 months
  variation in global longitudinal strain, diastolic parameters and degree of ventricular hypertrophy
cardiovascular outcomes | 24 months
  composite endpoint of death and heart failure hospitalization

SECONDARY OUTCOMES:
major cardiac arrhythmias | 24 months
  bradyarrhythmia, new-onset atrial fibrillation, ventricular tachycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No